CLINICAL TRIAL: NCT02905084
Title: Multi-physics Modeling the Physiology of a Patient in Critical Condition
Acronym: Physios
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-33
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Patient Care in ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The environment of the ICU and operating room allows the multi continuous monitoring of patients in critical situations. The physician anesthesiologist is working more and more in an environment where he receives a multitude of information from both the patient's medical history but also measured data in real time to its physiological situation. It is sometimes difficult for practitioners to consider all of the information by identifying a course of action. A decision support and a degree of automation can increase security along the lines of what has been observed in many processes and industries like aviation.

The goal of this project is to establish initially a database of physiological parameters. We want to use patient data to model physiological processes in order to advance towards the creation of "physios" program,

ELIGIBILITY:
Inclusion Criteria:

* Patient in intensive care unit ward

Exclusion Criteria:

* Patient or familly refusing participating to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in intensive care unit
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between high blood pressure measurement during the first 24h in ICU and number of patient alive at 28 days post ICU | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille; Salah BOUSSEN, MD, Principal Investigator — michelsalah.boussen@ap-hm.fr
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No